CLINICAL TRIAL: NCT06550505
Title: Evaluation and Follow-up of a Protocol for the Management of the Patient at High Risk Hemorrhagic in Cardiac Surgery by Monitoring Viscoelastic Hemostasis.
Brief Title: Management of the Patient at High Risk Hemorrhagic in Cardiac Surgery by Monitoring Viscoelastic Hemostasis.
Acronym: ELASTICC
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0017 - ELASTICC
Record Dates: First submitted 2021-11-30; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation and following of a protocol using viscoelastic test for the management of high risk patients in cardiac surgery

DETAILED DESCRIPTION:
Haemorragy is a frequent issue in cardiac surgery due to multiple contributing factors. Excessive bleeding as well as transfusion are associated with increased morbidity and mortality.

Haemostatic blood products (Fibrinogen, fresh frozen plasma, platelets) transfusion had historically been guided by routine coagulation tests (aPTT, PT, platelets and fibrinogen). However, the delay (Up to 60 minutes) often leads to an empirical use of blood products in a context where clinical judgment is unreliable due to the multiples mechanisms contributing to haemostatic failure.

Using viscoelastic tests (VET) in this context has several advantages :

* A quicker response (with first results from 10 minutes)
* An overall evaluation of haemostatic from the clot formation to its dissolution.

The use of VET has mainly been evaluated in cardiac surgery, with several recent meta-analysis : The use of transfusion algorithms based on VET is associated with less transfusions of red blood cell concentrates, plasma and platelets and also with less mortality, less re-interventions due to excessive bleeding and less post operative renal failure.

These data led the international society for the study of hemostasis and thrombosis (ISTH) to recommend their use of VET in cardiac surgery. In France, the proposals of the peri operative hemostatis group of interest (GIHP) also support their use, specifying that there is no unique consensual algorithm.

Considering this, the investigator established a transfusion algorithm based on the Quantra, a viscoelastic device using sonorrheometry, to guide transfusion in high-risk of bleeding cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria :

* Adult patients
* Elective or non-elective high risk of bleeding heart surgery
* Non-opposition

Exclusion Criteria:

* Pregnant women
* Age < 18 years
* Patients under guardianship
* Opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients. Elective or non-elective heart surgery. High risk of bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
fresh frozen plasma transfusion | 48 hours
  Proportion of patients transfused with fresh frozen plasma 48 hours after the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU BREST, Hôpital de la Cavale Blanche, Brest, France